CLINICAL TRIAL: NCT03636919
Title: CRD and mHealth for Pollen Allergy in Southern Europe. A Multicenter Observational Study
Brief Title: Component Resolved Diagnostics (CRD) and mHealth for Pollen Allergy In Southern Europe.
Acronym: IT-2020-MC
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-68
Record Dates: First submitted 2018-08-16; First posted 2018-08-17 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: patient with pollen allergic rhinitis patients will filled an e-BOOK included questionnaires of life
  Interventions: Other: e-BOOK

INTERVENTIONS:
Other: e-BOOK — Patients will filled an e (carnet) included the questionnaire includes the Control of Allergic Rhinitis and Asthma Test (CARAT)

SUMMARY:
Pollen allergic rhinitis is a very common condition whose symptomatic treatment is not always sufficient or satisfactory. The indication for allergic immunotherapy (IT) therefore often arises. The indication is based on the interrogation of the patient (chronology and severity of symptoms) and skin tests. But the interrogation, necessarily retrospective, brings often vague information and skin tests can be positive for allergens that have no clinical role (cross allergies).

The objective of the project is to help the clinician in the indication of the IT, on the one hand by setting up a prospective and computerized collection of symptoms by a computer logbook accessible by the mobile phone of the patient. on the other hand by performing on the patient's serum a molecular diagnosis allow the identification of the major allergens to which the patient is sensitized.

The same study will be conducted in 7 centers in southern European countries in patients aged 10 to 60 years with pollinosis. The examinations added by the research will take place during two routine visits: during a first visit, these patients will answer a standardized questionnaire, have a battery of allergological skin tests and a blood sample for molecular diagnosis. An application will then be loaded on their mobile phone and they will record their symptoms and medication during the pollen season. During a second visit, at the end of the pollen season, the allergist, in view of the data collected in the electronic notebook and the results of the molecular diagnosis will be able to prescribe a possible IT.

DETAILED DESCRIPTION:
Pollen allergic rhinitis is a very common condition whose symptomatic treatment is not always sufficient or satisfactory. The indication for allergic immunotherapy (IT) therefore often arises. The indication is based on the interrogation of the patient (chronology and severity of symptoms) and skin tests. But the interrogation, necessarily retrospective, brings often vague information and skin tests can be positive for allergens that have no clinical role (cross allergies).

The objective of the project is to help the clinician in the indication of the IT, on the one hand by setting up a prospective and computerized collection of symptoms by a computer logbook accessible by the mobile phone of the patient. on the other hand by performing on the patient's serum a molecular diagnosis allow the identification of the major allergens to which the patient is sensitized.

The same study will be conducted in 7 centers in southern European countries (where the diagnosis of pollen allergies is the most complex) in patients aged 10 to 60 years with pollinosis. The examinations added by the research will take place during two routine visits: during a first visit, these patients will answer a standardized questionnaire, have a battery of allergological skin tests and a blood sample for molecular diagnosis. An application will then be loaded on their mobile phone and they will record their symptoms and medication during the pollen season. During a second visit, at the end of the pollen season, the allergist, in view of the data collected in the electronic notebook and the results of the molecular diagnosis will be able to prescribe a possible IT.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18, good French, possession of a SmartPhone, Android or i-Phone, signature of the consent form.

Exclusion Criteria:

* Immunotherapy already performed, other severe chronic disease (eg dysimmunitary disease, immunodeficiency, chronic sinusitis and nasal polyposis), residence more than 30 km from the pollen sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting a Pollen allergic rhinitis
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
adapted treatment | 8 months
  The number of patients who had recourse to the theoretical treatment of AIT

CONTACTS AND LOCATIONS:
Overall Officials: emilie garrido pradalie, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France